CLINICAL TRIAL: NCT06837129
Title: Intravenous Nalbuphine for Prevention of Intrathecal Morphine-induced Nausea and Vomiting in Patients Undergoing Cesarean Section: A Double-blind, Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, PREEYAPHAN ARUNAKUL, Assistant Professor Preeyaphan Arunakul MD, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MTU-EC-AN-1-130/66
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Intrathecal Morphine; Caesarean Section; Postoperative Nausea and Vomiting; Neuraxial Opioid
Keywords: Postoperative Nausea and Vomiting; intrathecal morphine; caesarean section; neuraxial opioid
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV NALBUPHINE (Experimental): A single dose of 4 MG IV nalbuphine is given after cord clamping in study group
  Interventions: Drug: A single dose of 4 mg iv nalbuphine
- conventional (No Intervention): no medications is given

INTERVENTIONS:
Drug: A single dose of 4 mg iv nalbuphine — prevention of nausea vomiting
  Arms: IV NALBUPHINE

SUMMARY:
We study efficacy of iv nalbuphine in prevention of intrathecal morphine-induced nausea and vomiting in patients undergoing cesarean section.

DETAILED DESCRIPTION:
IV nalbuphine has been proved to help prevent intrathecal morphine-induced pruritus in some studies but results in nausea vomiting prevention have not been well studied. In Thailand, most caesarean section is done under spinal anesthesia with intrathecal morphine, proving that iv nalbuphine is effective would be beneficial for our population. This study aims to see whether 4 mg of nalbuphine is effective in reducing incidence of intrathecal morphine-related nausea vomiting in parturient who underwent C-section under spinal anesthesia with 0.2 mg of intrathecal morphine.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section under spinal anesthesia
* age > 18 years

Exclusion Criteria:

* Patients with known allergy to medications used in this study (nalbuphine, bupivacaine or morphine)
* Patient with medical conditions which spinal anesthesia is contraindicated ie. heart diseases, renal or hepatic impairment, obesity >=100 kilograms
* Patients with history of postoperative nausea and vomiting (PONV) or motion sickness who may have preexisting risk factors for PONV
* Patient with known history of drug abuse
* Unwilling to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea vomiting in 24 hours | 24 hours

SECONDARY OUTCOMES:
Severity of nausea vomiting | 24 hours
Postoperative pain score | 24 hours
Incidence of pruritus | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Assist. Prof. Dr. Preeyaphan Arunakul, M.D., FRCAT, Principal Investigator — Thammasat University
Locations (2):
- Thailand (2):
  - Department of Anesthesiology, Faculty of Medicine, Thammasat University, Pathum Thani, Changwat Pathum Thani
  - Faculty of Medicine Thammasat University, Pathum Thani, Changwat Pathum Thani

IPD SHARING:
Plan to Share IPD: No